CLINICAL TRIAL: NCT00457886
Title: Serum Levels of Hormones Known to Affect Parturition in Patients Receiving 17 Alpha-Hydroxyprogesterone Caproate (17-P) for the Prevention of Preterm Delivery
Brief Title: Measurement of Hormone Levels in Patients Receiving 17-HPC for Preterm Delivery
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: Wedgewood Pharmacy (Industry); National Center for Research Resources (NCRR) (NIH)
Other Study IDs: IRB 2005-142
Record Dates: First submitted 2007-04-06; First posted 2007-04-09 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Preterm Delivery
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to measure hormones in the blood known to affect the timing of delivery after a single injection of 17-P in order to help understand its mechanism of action in preventing preterm delivery.

DETAILED DESCRIPTION:
A recent study by Meis and colleagues published in the New England Journal of Medicine in June 2003 demonstrated a 33% reduction in the rate of preterm delivery in patients with a previous history of preterm delivery who then used weekly 17-P injections in the subsequent pregnancy.

This is a milestone in the prevention of preterm delivery and is the reason you have chosen to receive treatment with 17-P.

However, how 17-P works to prevent preterm delivery is unclear. Knowledge of the mechanism of action of 17-P would help in selecting patients for treatment and may be useful in monitoring the efficacy of therapy.

Studies have suggested that the timing of delivery depends on a type of placental clock, affected by levels of corticotropin-releasing hormone (CRH) and progesterone (P).

CRH can be thought to act as an accelerator, and P as a brake. Serial injections of 17-P beginning in the second trimester of pregnancy may prevent preterm delivery by maintaining progesterone dominance, and be reflected in increased levels of progesterone and/or 17-P, or decreased levels of cortisol and/or CRH. These are the hormones that will be measured in this study.

Results of the study will be important whatever the outcome. If there is no measurable change in the hormones measured, this is important to know and investigation of other markers can be pursued. If there is a measurable change in the hormones measured, then this pilot study could serve to support a larger more definitive study, which could lead to very valuable information relating to the practical use of 17-P for the prevention of preterm delivery.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous preterm delivery in a previous pregnancy, are between 15-20 weeks gestation during the current pregnancy, and have already decided whether or not to receive 17-alphahydroxyprogesterone caproate (17-P) for the prevention of preterm delivery.

Exclusion Criteria:

* Multiple gestation
* Known fetal anomaly
* Progesterone or heparin treatment during the current pregnancy
* Seizure disorder
* Pre-existing or gestational diabetes
* Hypertension requiring medication
* Thyroid or adrenal gland disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 20
Dates: Start 2005-07; Study Completion 2007-06

CONTACTS AND LOCATIONS:
Overall Officials: John Queenan, MD, Study Director — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States